CLINICAL TRIAL: NCT01435980
Title: Study of Comparison the Treatment Effect Between Gastric Bypass and Exenatide in Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wu Qinan (Other)
Responsible Party: Sponsor-Investigator, Wu Qinan, Third Military Medical University, Third Military Medical University
Organization: Third Military Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: the south west Hospital2
Record Dates: First submitted 2011-09-08; First posted 2011-09-19 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; Gastric Bypass; GLP-1; adiponectin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gastric Bypass; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- basal treatment (No Intervention): basal treatment
- Gastric Bypass (Experimental): basal treatment and Gastric Bypass
  Interventions: Procedure: Gastric Bypass
- Exenatide (Experimental): basal treatment and Exenatide
  Interventions: Drug: Exenatide

INTERVENTIONS:
Procedure: Gastric Bypass — basal treatment and Gastric Bypass
  Other Names: basal treatment + Gastric Bypass
  Arms: Gastric Bypass
Drug: Exenatide — basal treatment and Exenatide
  Other Names: basal treatment + Exenatide
  Arms: Exenatide

SUMMARY:
Objectives: To investigate the treatment effect between Gastric Bypass and Exenatide in Type 2 Diabetes in our hospital, in order to investigate the possible mechanism of Gastric Bypass and Exenatide.

DETAILED DESCRIPTION:
Methods:

60 Type 2 diabetes in our hospital will divide into 3 groups: group A (20 patients who give basal treatment), group B (20 patients who give basal and Exenatide treatment, group C（20 patients who give basal and Gastric Bypass treatment). The age, height, weight, blood glucose, glycosylated hemoglobin A1c（HbA1c）,homeostasis model assessment(HOMA-IR), lipid, blood pressure, course of disease, ejection fraction (EF), fractional shortening(FS), diameter of left ventricle in late diastolic stage(LVEDd), the thickness of the ventricular septa（IVSD) and the posterior wall of the right ventricle in late diastolic stage (LVPWd) will record respectively. Left ventricular mass index (LVMI), relative wall thickness (RWT) will calculate and High-sensitive C-reactive protein (HsCRP), adiponectin and Tumor necrosis factor-α（TNF-α） will detect as Baseline. After each group's treatment, Change from baseline of all indexes will record, Multifactor logistic regression will be analyzed the correlations between each positive indexes.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥ 35kg/m2, With Type 2 Diabetes;
2. BMI32-34.9kg/m2, With Type 2 Diabetes, Insulin Therapy in Combination With Oral Administration of Drugs for 6 Months and HbA1c ≥ 7%;
3. Between the Ages of 18-60 Years;
4. Course of Type 2 Diabetes ≤ 5 Years;
5. ICA, IAA, GAD Are Negative , C-peptide Level is Not Less Than 0.3mg / L;

Exclusion Criteria:

1. non-diabetic patients , type 1 diabetes (serum insulin antibodies (ICA) or glutamic acid decarboxylase antibodies (GADA)-positive autoimmune diabetes), special type of diabetes, gestational diabetes;
2. patients who had liver or renal failure
3. severe infections in patients and patients who had cerebrovascular disease
4. patients who had heart failure
5. fasting serum insulin or 2-hour postprandial serum insulin were lower than normal (<20mmol / L)
6. course of diabetes> 5 years or age> 60 years or age <18 years

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-02; Primary Completion 2016-01 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Clinical events | 1 year
  Participant with stroke or Myocardial infarction or acute diabetic complication or Liver and renal failure or death or other Adverse Events.

SECONDARY OUTCOMES:
echocardiography | 1 year
  Left ventricular mass index (LVMI)
echocardiography | 1 year
  relative wall thickness (RWT)
Blood testing | 1 year
  High-sensitive C-reactive protein (HsCRP)
Blood testing | 1 year
  homeostasis model assessment(HOMA-IR)
Blood testing | 1 year
  adiponectin
Blood pressure monitoring | 1 month
  blood pressure
Blood testing | 1 year
  glycosylated hemoglobin A1c（HbA1c）

CONTACTS AND LOCATIONS:
Overall Officials: liang zi wen, doctor, Principal Investigator — Third Military Medical University
Locations (1):
- Endocrine Department, the south west Hospital of the Third Military Medical University, Chongqing, Chongqing Municipality, China